CLINICAL TRIAL: NCT06617182
Title: Efficacy and Safety of Thalidomide Combined With Glutamine in the Treatment of Radiation Intestinal Injury: a Single-center, Open-label, Randomized Controlled Study
Brief Title: Efficacy and Safety of Thalidomide Combined With Glutamine in the Treatment of Radiation Intestinal Injury.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yongquan Shi (Other)
Responsible Party: Sponsor-Investigator, Yongquan Shi, Professor, Xijing Hospital of Digestive Diseases
Organization: Xijing Hospital of Digestive Diseases (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20242229-F-1
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Radiation Enteritis
MeSH Terms: interventions — Thalidomide; Glutamine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The thalidomide group (Experimental): Patients in the thalidomide group will receive oral thalidomide at a dosage of 100 mg one time daily for 8 weeks.
  Interventions: Drug: Thalidomide
- The glutamine group (Experimental): Patients in the glutamine group were given two enteric-soluble capsules of compound glutamine three times a day for 8 weeks.
  Interventions: Drug: Glutamine
- The thalidomide combined with glutamine group (Experimental): Patients in the thalidomide combined with glutamine group will receive oral thalidomide at a dosage of 100 mg one time daily and two enteric-soluble capsules of compound glutamine three times a day for 8 weeks.
  Interventions: Drug: Thalidomide+Glutamine

INTERVENTIONS:
Drug: Thalidomide — Patients in thalidomide group took thalidomide orally at a dose of 100mg once a day for 8 weeks.
  Arms: The thalidomide group
Drug: Glutamine — In the glutamine group, two capsules of glutamine were taken orally 3 times a day for 8 weeks.
  Other Names: Compound glutamine enteric-coated capsules
  Arms: The glutamine group
Drug: Thalidomide+Glutamine — Patients in thalidomide combined with glutamine group took thalidomide orally at a dose of 100mg once a day and two capsules of glutamine were taken orally 3 times a day for 8 weeks.
  Arms: The thalidomide combined with glutamine group

SUMMARY:
At present, there is still a lack of standard and effective treatment strategies and procedures for radiation intestinal injury. Studies have shown that thalidomide can effectively treat refractory gastrointestinal bleeding caused by vascular malformation. Therefore, The investigators designed a single-center, open-label, randomized controlled study to evaluate the efficacy and safety of thalidomide combined with glutamine in the treatment of radiation intestinal injury.

DETAILED DESCRIPTION:
Screening: This phase will not last longer than one week, and the subject will be assessed for eligibility after signing the informed consent form.

Treatment: Subjects were randomly assigned to three different treatment groups for 8 weeks.

Follow-up: The subjects' defecation status was recorded every day during treatment, telephone follow-up was conducted every two weeks, and laboratory indicators (including blood routine, stool routine, etc.) were tested every four weeks. The test was terminated one week after treatment and the improvement of subjects' stool blood was assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old, gender is not limited;
* Patients with hematochezia symptoms of chronic radiation intestinal injury: Due to the lack of diagnostic gold standard for radiation intestinal injury, a comprehensive analysis of clinical, endoscopic, imaging and histopathological findings was mainly performed to make the diagnosis of radiation intestinal injury on the basis of excluding infectious and other non-infectious intestinal injuries. Exposure to radioactive sources is a necessary factor in the diagnosis of radiation intestinal injury, and tumor activity or recurrence should be excluded.
* The proportion of dominant defecation bleeding in total defecation times in the week before treatment is not less than 20%;
* ECOG score: 0-2.

Exclusion Criteria:

* Patients with hemodynamic instability;
* Patients with obvious liver and kidney function injury: bilirubin, aminotransferase (ALT, AST) exceeded the upper limit of normal by 2 times; eGFR<60ml/min or dialysis patients;
* Patients allergic to thalidomide or glutamine;
* Patients whose primary disease was gastrointestinal malignancy;
* Patients currently suffering from serious or uncontrolled underlying diseases of the blood, digestive tract, metabolism, endocrine, lung, heart, nervous system, mental system, etc.;
* Female patients during pregnancy and breastfeeding (including patients with reproductive needs);
* Patients infected with HIV;
* Patients who cannot cooperate with regular follow-up and review of laboratory indicators;
* any other circumstances which, in the opinion of the investigator, would render the subject unfit for study inclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Treatment response rate. | From enrollment to the end of treatment at 8 weeks.
  The proportion of overt defecation bleeding in total defecation within 1 week after treatment was reduced by ≥50% compared with 1 week before treatment.

SECONDARY OUTCOMES:
No further bleeding occurred within 1 week after treatment | From enrollment to the end of treatment at 8 weeks.
  Stool occult blood negative 2 times in a row on different dates
Number of blood transfusions during the treatment period | From enrollment to the end of treatment at 8 weeks.
  times
Red blood cell input | From enrollment to the end of treatment at 8 weeks.
  Input red blood cells according to the situation
Hemoglobin level | From enrollment to the end of treatment at 8 weeks.
  Record each test result
Number of hospitalizations due to bleeding | From enrollment to the end of treatment at 8 weeks.
  times
Number of days in hospital due to bleeding | From enrollment to the end of treatment at 8 weeks.
  days
Require surgery | From enrollment to the end of treatment at 8 weeks.
  yes or no

IPD SHARING:
Plan to Share IPD: No